CLINICAL TRIAL: NCT00137020
Title: A Multi-Center Study to Examine The Clinical Effects of Cross Titration of Antipsychotics With Ziprasidone in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: Clinical Effect Of Cross Titration Of Antipsychotics With Ziprasidone In Schizophrenia Or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281117
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia; Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone

INTERVENTIONS:
Drug: ziprasidone

SUMMARY:
The primary objective is to compare effectiveness of ziprasidone treatment to current treatments (haloperidol, olanzapine or risperidone) measured by change in Brief Psychiatric Rating Scale (BPRS) scores versus baseline

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of schizophrenia or schizoaffective disorder, using DSM-IV criteria.
* Currently receiving either haloperidol, olanzapine or risperidone within -/+ 25% of the recommended daily dose (as delineated by the medication's package insert

Exclusion Criteria:

* Resistance to conventional antipsychotic drugs
* With antipsychotic agents other than olanzapine, risperidone or haloperidol at start of treatment regimen within 12 hours prior to first dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294
Dates: Start 2004-11; Study Completion 2006-04

PRIMARY OUTCOMES:
The primary efficacy variable will be change from baseline in Brief Psychiatric Rating Scale (BPRS) total score

SECONDARY OUTCOMES:
Change From Baseline In Clinical Global Impression Severity (CGI-S)
Clinical Global Impression Improvement (CGI-I)
Change From Baseline In Positive and Negative Syndrome Scale (PANSS) Total
Change from baseline in scores on the Montgomery-Asberg Depression Rating Scale (MADRS)
Change from baseline in scores on the MADRS Without Items 4, 5
Change from baseline in Global Assessment of Functioning (GAF)
Change From Baseline In Drug Attitude Inventory (DAI)
Change From Baseline In Weight
Change From Baseline In Prolactin And Lipid Levels
Change From Baseline in Modified Simpson Angus Scale (m-SAS) Total Score
Change From Baseline in Barnes Akathisia Scale (BAS)
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS)- Movement Ratings Total Score
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS)- Global Judgment Of Severity Total Score

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- Egypt (4):
  - Pfizer Investigational Site, Alexandria
  - Pfizer Investigational Site, Asyut
  - Pfizer Investigational Site, Cairo
  - Pfizer Investigational Site, Tanta
- Greece (2):
  - Pfizer Investigational Site, Larissa, Mezourlo
  - Pfizer Investigational Site, Athens
- Pfizer Investigational Site, Jordan, Jordan
- Pfizer Investigational Site, Kuwait City, Kuwait
- Pfizer Investigational Site, Beirut, Lebanon
- Pfizer Investigational Site, Khobar, Saudi Arabia
- South Africa (6):
  - Pfizer Investigational Site, Garankuwa, Gauteng
  - Pfizer Investigational Site, Krugersdorp, Gauteng
  - Pfizer Investigational Site, Noordheuwel, Krugersdorp, Gauteng
  - Pfizer Investigational Site, Bellair, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Pinetown, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Observatory, Cape Town, Western Cape
- Turkey (Türkiye) (7):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Bursa
  - Pfizer Investigational Site, Erzurum
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir
  - Pfizer Investigational Site, Manisa
  - Pfizer Investigational Site, Şişli
- Pfizer Investigational Site, Dubai, United Arab Emirates

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281117&StudyName=Clinical+Effect+Of+Cross+Titration+Of+Antipsychotics+With+Ziprasidone+In+Schizophrenia+Or+Schizioaffective+Disorder